CLINICAL TRIAL: NCT04524663
Title: A Phase 2 Randomized, Double Blinded, Placebo Controlled Study of Oral Camostat Mesilate Compared to Standard of Care in Subjects With Mild-Moderate COVID-19
Brief Title: Oral Camostat Compared With Standard Supportive Care in Mild-Moderate COVID-19 Patients
Acronym: COPS-2003
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 56029
Record Dates: First submitted 2020-04-10; First posted 2020-08-24 (Actual); Results first posted 2022-06-10 (Actual); Last update posted 2022-06-10 (Actual); Status verified 2022-06

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19 | interventions — camostat

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Camostat mesilate (Experimental): Patients will receive camostat mesilate for 10 days in addition to standard of care treatment.
  Interventions: Drug: Camostat Mesilate; Other: Standard of Care Treatment
- Placebo (Placebo Comparator): Study participants will receive placebo to match camostat mesilate for 10 days in addition to standard of care treatment.
  Interventions: Drug: Placebo; Other: Standard of Care Treatment

INTERVENTIONS:
Drug: Camostat Mesilate — Camostat Mesilate administered as oral tablets
  Other Names: Foipan®
  Arms: Camostat mesilate
Drug: Placebo — Placebo to match camostat mesilate
  Arms: Placebo
Other: Standard of Care Treatment — Standard of Care Treatment for COVID-19 Infection

SUMMARY:
This study will evaluate the efficacy of oral Foipan® (camostat mesilate) compared with the current standard of care in reducing the duration of viral shedding of SARS-CoV-2 virus in patients with mild-moderate COVID-19 disease.

Patients will attend 4 study visits over a period of up to 28 days.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of COVID-19 disease as presence of mild-moderate symptoms without signs of respiratory distress, with FDA-cleared molecular diagnostic assay positive for SARS-CoV-2 within 72 hours prior to informed consent
* Males must be sterile, OR agree not to donate semen AND agree to strictly adhere to contraceptive measures during the study and for seven days following the last dose of study medication
* Females must be unable to bear children, OR ensure that their male partner is incapable of fathering a child, OR, if of childbearing potential will strictly adhere to contraceptive measures during the study and for seven days following the last dose of study medication
* Females must agree to stop breast-feeding prior to first dose of study drug and through seven days after completing therapy
* Females must have a negative pregnancy test at screening
* Participant agrees to maintain home or other quarantine as recommended by the study physician, except to visit the study site as required by the protocol

Exclusion Criteria:

* Concomitant bacterial respiratory infection documented by respiratory culture. NOTE: Subjects on empirical antibiotic treatment for possible but unproven bacterial pneumonia, but who are positive for SARS-CoV-2, are allowed in the study.
* Previous use of antiviral drugs that may be active against Covid-19.
* Abnormal laboratory test results at screening:
* Use of adrenocorticosteroids (except topical or inhaled preparations or oral preparations equivalent to or less than 10 mg of oral prednisone) or immunosuppressive or immunomodulatory drugs (e.g., immunosuppressants, anticancer drugs, interleukins, interleukin antagonists or interleukin receptor blockers). NOTE: Treatment of study participants following institutional COVID-19 treatment policies or guidelines, including the use of immunomodulatory medications, is permitted. This excludes treatment with agents that have the potential for direct antiviral activity, including convalescent plasma and NO, and co-enrollment into other clinical studies that evaluate investigational agents for COVID-19.
* Serious chronic disease (e.g., human immunodeficiency virus [HIV], cancer requiring chemotherapy within the preceding 6 months, and/or moderate or severe hepatic insufficiency).
* Previously received camostat mesilate within the past 30 days.
* Advanced kidney disease
* Advanced liver disease
* History of alcohol or drug abuse in the previous 6 months.
* Psychiatric illness that is not well controlled (defined as stable on a regimen for more than one year).
* Taken another investigational drug within the past 30 days.
* Seemed by the Investigator to be ineligible for any reason.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2020-12-19 (Actual); Primary Completion 2021-05-15 (Actual); Study Completion 2021-05-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julie Parsonnet, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: After 49 participants were enrolled, this trial was subsumed into a pragmatic platform trial (the COVID-19 Outpatient Pragmatic Platform Study (COPPS) - Camostat Sub-Protocol (NCT04662073). Additional subjects subsequently consented for camostat in the platform study. Their results are not included here.
Groups:
- Camostat Mesilate: Camostat mesilate for 10 days in addition to standard of care treatment.
- Placebo: Placebo to match camostat mesilate for 10 days in addition to standard of care treatment.
Period: Overall Study
Arm/Group | Camostat Mesilate | Placebo
Started | 25 | 24
Completed | 25 | 22
Not Completed | 0 | 2
Not completed — Withdrawal by Subject | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Camostat Mesilate | Placebo | Total
Number analyzed (Participants) | 25 | 24 | 49
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.88 (13.47) | 40.54 (14.27) | 39.18 (13.79)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 7 | 17
  Male | 15 | 17 | 32
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Patient selected one of the options in a survey. Ethnicity was an optional survey item. Population: Participants who provided ethnicity data are included in the analysis.
  Participants
    number analyzed (Participants) | 24 | 22 | 46
    Hispanic or Latino | 6 | 9 | 15
    Not Hispanic or Latino | 18 | 13 | 31
    Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Patient selected one of the options in a survey. Race was an optional survey item. Population: Participants who provided race data are included in the analysis.
  Participants
    American Indian/Alaska Native: number analyzed (Participants) | 23 | 18 | 41
    American Indian/Alaska Native | 1 | 0 | 1
    Asian: number analyzed (Participants) | 23 | 18 | 41
    Asian | 5 | 4 | 9
    Native Hawaiian or other Pacific Islander: number analyzed (Participants) | 23 | 18 | 41
    Native Hawaiian or other Pacific Islander | 1 | 0 | 1
    Black or African American: number analyzed (Participants) | 23 | 18 | 41
    Black or African American | 1 | 0 | 1
    White: number analyzed (Participants) | 23 | 18 | 41
    White | 12 | 7 | 19
    More than one race: number analyzed (Participants) | 23 | 18 | 41
    More than one race | 0 | 1 | 1
    Unknown: number analyzed (Participants) | 23 | 18 | 41
    Unknown | 1 | 0 | 1
    Other: number analyzed (Participants) | 23 | 18 | 41
    Other | 2 | 6 | 8
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 25 | 24 | 49
Anterior nares RT-PCR Ct [Median (Inter-Quartile Range); unit: cycles] — Cycle threshold (Ct) denotes how many PCR cycles are required before the SARS-CoV-2 viral RNA reached a detectable level. Higher Ct values correspond to lower viral copy numbers. For reference, Ct values of 20 correspond to ~2.12 x 106 viral copies per milliliter, while a Ct value of 40 is undetectable and is considered the lower limit of detection of this RT-PCR test for SARS-CoV-2. RT-PCR: reverse transcription-polymerase chain reaction. Population: Participants with baseline data are included in the analysis.
  cycles
    number analyzed (Participants) | 20 | 22 | 42
    (all) | 19.40 [17.17 to 24.40] | 21.58 [17.98 to 26.84] | 20.87 [17.33 to 25.06]
Duration of Symptoms [Median (Inter-Quartile Range); unit: days] — Population: Participants with baseline data are included in the analysis.
  days
    number analyzed (Participants) | 24 | 24 | 48
    (all) | 5.00 [2.75 to 6.00] | 4.50 [3.75 to 5.00] | 5.00 [3.00 to 6.00]
Number of Symptoms [Median (Inter-Quartile Range); unit: symptoms] | 6 [3 to 7] | 6 [4 to 8] | 6 [3 to 8]
Body Mass Index [Median (Inter-Quartile Range); unit: kg/m^2] | 27.81 [24.89 to 33.36] | 28.00 [24.97 to 30.15] | 27.81 [24.89 to 32.09]
Aspartate Aminotransferase [Median (Inter-Quartile Range); unit: units/L] | 25.00 [21.00 to 29.00] | 30.00 [24.75 to 35.00] | 27.00 [22.00 to 35.00]
Alanine Aminotransferase [Median (Inter-Quartile Range); unit: units/L] | 25.00 [20.00 to 35.00] | 34.50 [20.00 to 48.50] | 29.00 [20.00 to 44.50]
Uric acid [Median (Inter-Quartile Range); unit: mg/dL] — Population: Participants with baseline data are included in the analysis.
  mg/dL
    number analyzed (Participants) | 23 | 24 | 47
    (all) | 5.10 [4.40 to 5.85] | 5.00 [3.88 to 5.85] | 5.10 [4.05 to 5.85]
Creatinine [Median (Inter-Quartile Range); unit: mg/dL] | 0.87 [0.68 to 0.97] | 0.86 [0.67 to 0.98] | 0.87 [0.68 to 0.98]

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Curve (AUC) of Shedding of SARS-CoV-2 Virus
Description: AUC of shedding of SARS-CoV-2 virus calculated using the reverse transcription-polymerase chain reaction (RT-PCR) measures of viral load from self-collected nasal swabs on days 1-10. AUC was defined by a single participant's cycle threshold (Ct) from nasal swabs collected and calculated by the trapezoidal rule, using exact times of collection of each swab. Ct denotes how many PCR cycles are required before the SARS-CoV-2 viral RNA reached a detectable level. Higher Ct values correspond to lower viral copy numbers. For reference, Ct values of 20 correspond to ~2.12 x 106 viral copies per milliliter, while a Ct value of 40 is undetectable and is considered the lower limit of detection of this RT-PCR test for SARS-CoV-2.
Time Frame: Days 1-10
Population: Patients with nasal swab data are included in the analysis.
Measure: Median (Inter-Quartile Range); unit: cycles*days
Arm/Group | Camostat Mesilate | Placebo
Number analyzed (Participants) | 22 | 24
cycles*days | 95.3 [66.7 to 124] | 93 [68 to 124]
Statistical Analysis 1: Comparison: Camostat Mesilate vs Placebo; Test type: Superiority; p = 0.89, Regression, Linear; Median Difference (Net) = 0.59, 95% CI 2-sided [-8.14 to 9.32]

2. Secondary Outcome: AUC of Shedding of SARS-CoV-2 Virus
Description: AUC of shedding of SARS-CoV-2 virus calculated using the RT-PCR measures of viral load from self-collected nasal swabs on days 1-10, 14, 21, and 28. AUC was defined by a single participant's Ct from nasal swabs collected and calculated by the trapezoidal rule, using exact times of collection of each swab. Ct denotes how many PCR cycles are required before the SARS-CoV-2 viral RNA reached a detectable level. Higher Ct values correspond to lower viral copy numbers. For reference, Ct values of 20 correspond to ~2.12 x 106 viral copies per milliliter, while a Ct value of 40 is undetectable and is considered the lower limit of detection of this RT-PCR test for SARS-CoV-2.
Time Frame: Days 1-10, 14, 21, and 28
Population: Patients with nasal swab data are included in the analysis.
Measure: Median (Inter-Quartile Range); unit: cycles*days
Arm/Group | Camostat Mesilate | Placebo
Number analyzed (Participants) | 22 | 24
cycles*days | 116 [68.7 to 157] | 124 [71.8 to 169]
Statistical Analysis 1: Comparison: Camostat Mesilate vs Placebo; Test type: Superiority; p = 0.02, Regression, Linear; Median Difference (Net) = 18.9, 95% CI 2-sided [2.98 to 34.83]

3. Secondary Outcome: Time Until Cessation of Shedding of SARS-CoV-2 Virus
Description: This outcome is defined as the time in days from randomization to the first negative RT-PCR result of self-collected nasal swabs that is followed by only negative results (i.e. no later positive results are observed).
Time Frame: Up to 28 days
Population: Patients with nasal swab data are included in the analysis.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Camostat Mesilate | Placebo
Number analyzed (Participants) | 22 | 24
days | 14 [7 to 21] | 21 [12 to NA] — Not estimable (curve did not reach the 75th percentile)
Statistical Analysis 1: Comparison: Camostat Mesilate vs Placebo; Test type: Superiority; p = 0.24, Cox proportional hazards model; Hazard Ratio (HR) = 1.69, 95% CI 2-sided [0.70 to 4.10]

4. Secondary Outcome: Clinical Worsening of COVID-19 Disease in Symptomatic Patients
Description: Number of symptomatic patients with clinical worsening, defined as the development of respiratory distress or symptoms that require hospitalization.
Time Frame: Up to 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Camostat Mesilate | Placebo
Number analyzed (Participants) | 25 | 24
Participants | 2 | 0
Statistical Analysis 1: Comparison: Camostat Mesilate vs Placebo; Test type: Superiority; p = 0.49, Fisher Exact

5. Secondary Outcome: Time Until Resolution of Symptoms
Description: This outcome is defined as absence of moderate or severe symptoms for at least 24 hours for those reporting moderate or severe symptoms at baseline.
Time Frame: Up to 28 days
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Camostat Mesilate | Placebo
Number analyzed (Participants) | 25 | 24
days | 11 [5 to 16] | 12 [9 to NA] — Not estimable (curve did not reach the 75th percentile)
Statistical Analysis 1: Comparison: Camostat Mesilate vs Placebo; Test type: Superiority; p = 0.24, Cox proportional hazards model; Hazard Ratio (HR) = 0.65, 95% CI 2-sided [0.32 to 1.33]

6. Secondary Outcome: Development of Antibodies to SARS-CoV-2
Description: Number of patients that develop antibodies to SARS-CoV-2.
Time Frame: Up to 28 days
Population: Data were not collected for this outcome measure.
Arm/Group | Camostat Mesilate | Placebo
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Drug Level on Day Five, One Hour After a Dose Taken on an Empty Stomach
Time Frame: Day 5, 1 hour post dose
Population: Data were not collected for this outcome measure.
Arm/Group | Camostat Mesilate | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 28 days
Arm/Group | Camostat Mesilate | Placebo
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/25 | 3/24
Other Adverse Events (participants affected / at risk) | 2/25 | 10/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Camostat Mesilate (N=25) | Placebo (N=24)
Liver function tests (Investigations) | 0 | 1
Hypotension (Vascular disorders) | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Suidical ideation (Psychiatric disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Camostat Mesilate (N=25) | Placebo (N=24)
Liver function test (LFT) elevation (Investigations) | 1 | 4
Diarrhea (Gastrointestinal disorders) | 1 | 2
Rash (Skin and subcutaneous tissue disorders) | 0 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-12-04): https://cdn.clinicaltrials.gov/large-docs/63/NCT04524663/Prot_SAP_000.pdf